CLINICAL TRIAL: NCT00000513
Title: Trial of Antihypertensive Intervention Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 32; R01HL030171-05 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Reducing; Diet, Sodium-Restricted; Chlorthalidone; Atenolol

INTERVENTIONS:
Behavioral: diet, reducing
Behavioral: diet, sodium-restricted
Drug: chlorthalidone
Drug: atenolol

SUMMARY:
The objective of the Trial of Antihypertensive Intervention Management (TAIM) was to determine the efficacy of dietary management and/or drug therapy, namely thiazide-like diuretics or a beta-blocker, in the control of mild hypertension. Additionally, the Continuation of the Trial of Antihypertensive Intervention Management (COTAIM) tested the effects of long-term weight reduction, and sodium/potassium changes added to weight reduction, as well as the original drug treatment, on the failure rate of blood pressure control.

DETAILED DESCRIPTION:
BACKGROUND:

The Trial of Antihypertensive Intervention Management was an extension of the NHLBI-supported Dietary Intervention Study of Hypertension (DISH) which concluded in March 1984 and showed that either weight reduction or sodium restriction diets reduced relapse rates of hypertensives who had received long-term drug treatment and then been withdrawn from drugs. TAIM was initiated in April 1984 and continued for four years at three centers and added to DISH the art of evaluating combined drug and dietary treatments. COTAIM was continued at three clinical sites in July 1988. Analysis of COTAIM results continued through November 1994 under grant R01HL40072.

DESIGN NARRATIVE:

TAIM patients were randomly assigned to one of three diets and to one of three drug regimens. The dietary interventions consisted of a weight loss program, sodium reduction with increased potassium intake, or no change in diet. The drug regimen consisted of a beta-blocker (atenolol), a thiazide-like diuretic (chlorthalidone), or placebo. The major endpoint was change in diastolic blood pressure after six months of intervention. Individuals who did not reach goal blood pressure after six months received additional drugs. Other endpoints included total risk factor score change, psychological function, and lifestyle change.

COTAIM consisted of two studies with a total of 600 subjects. COTAIM I compared the TAIM weight loss group to a randomly selected half of the usual diet group. The primary endpoint of COTAIM I was the degree of control of blood pressure on initial TAIM therapy between TAIM baseline and the end of COTAIM, a five year period.

COTAIM II added a weight loss regimen both to the sodium restriction/potassium supplementation groups and to the other half of the usual diet group. The primary outcome was control of blood pressure on initial TAIM therapy between COTAIM baseline and the end of COTAIM, a two-year period.

ELIGIBILITY:
Men and women, ages 21 to 65, with mild hypertension in the range of 90 to 100 mm Hg diastolic blood pressure.

Subjects were obese (110-150 percent of ideal weight).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1984-04; Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morton Blaufox — Albert Einstein College of Medicine; Kent Kirchner — University of Mississippi Medical Center; Albert Oberman — University of Alabama at Birmingham; Sylvia Wassertheil-Smoller — Albert Einstein College of Medicine

REFERENCES:
- [Background] Davis BR, Blaufox MD, Hawkins CM, Langford HG, Oberman A, Swencionis C, Wassertheil-Smoller S, Wylie-Rosett J, Zimbaldi N. Trial of antihypertensive interventions and management. Design, methods, and selected baseline results. Control Clin Trials. 1989 Mar;10(1):11-30. doi: 10.1016/0197-2456(89)90016-0. PMID 2649308
- [Background] Langford HG, Rockhold RW, Wassertheil-Smoller S, Oberman A, Davis BR, Blaufox MD. Effect of weight loss on thiazide produced erectile problems in men. Trans Am Clin Climatol Assoc. 1990;101:190-4. PMID 2486442
- [Background] Oberman A, Wassertheil-Smoller S, Langford HG, Blaufox MD, Davis BR, Blaszkowski T, Zimbaldi N, Hawkins CM. Pharmacologic and nutritional treatment of mild hypertension: changes in cardiovascular risk status. Ann Intern Med. 1990 Jan 15;112(2):89-95. doi: 10.7326/0003-4819-112-2-89. PMID 1967210
- [Background] Langford HG, Davis BR, Blaufox D, Oberman A, Wassertheil-Smoller S, Hawkins M, Zimbaldi N. Effect of drug and diet treatment of mild hypertension on diastolic blood pressure. The TAIM Research Group. Hypertension. 1991 Feb;17(2):210-7. doi: 10.1161/01.hyp.17.2.210. PMID 1671380
- [Background] Wassertheil-Smoller S, Blaufox MD, Oberman A, Davis BR, Swencionis C, Knerr MO, Hawkins CM, Langford HG. Effect of antihypertensives on sexual function and quality of life: the TAIM Study. Ann Intern Med. 1991 Apr 15;114(8):613-20. doi: 10.7326/0003-4819-114-8-613. PMID 2003706
- [Background] Langford HG. Sodium-potassium interaction in hypertension and hypertensive cardiovascular disease. Hypertension. 1991 Jan;17(1 Suppl):I155-7. doi: 10.1161/01.hyp.17.1_suppl.i155. PMID 1986994
- [Background] Wassertheil-Smoller S, Blaufox MD, Oberman AS, Langford HG, Davis BR, Wylie-Rosett J. The Trial of Antihypertensive Interventions and Management (TAIM) study. Adequate weight loss, alone and combined with drug therapy in the treatment of mild hypertension. Arch Intern Med. 1992 Jan;152(1):131-6. PMID 1728908
- [Background] Davis BR, Oberman A, Blaufox MD, Wassertheil-Smoller S, Hawkins CM, Cutler JA, Zimbaldi N, Langford HG. Effect of antihypertensive therapy on weight loss. The Trial of Antihypertensive Interventions and Management Research Group. Hypertension. 1992 Apr;19(4):393-9. doi: 10.1161/01.hyp.19.4.393. PMID 1555871
- [Background] Wassertheil-Smoller S, Oberman A, Blaufox MD, Davis B, Langford H. The Trial of Antihypertensive Interventions and Management (TAIM) Study. Final results with regard to blood pressure, cardiovascular risk, and quality of life. Am J Hypertens. 1992 Jan;5(1):37-44. doi: 10.1093/ajh/5.1.37. PMID 1736933
- [Background] Blaufox MD, Lee HB, Davis B, Oberman A, Wassertheil-Smoller S, Langford H. Renin predicts diastolic blood pressure response to nonpharmacologic and pharmacologic therapy. JAMA. 1992 Mar 4;267(9):1221-5. PMID 1538559
- [Background] Davis BR, Blaufox MD, Oberman A, Wassertheil-Smoller S, Zimbaldi N, Cutler JA, Kirchner K, Langford HG. Reduction in long-term antihypertensive medication requirements. Effects of weight reduction by dietary intervention in overweight persons with mild hypertension. Arch Intern Med. 1993 Aug 9;153(15):1773-82. doi: 10.1001/archinte.153.15.1773. PMID 8333814
- [Background] Wylie-Rosett J, Wassertheil-Smoller S, Blaufox MD, Davis BR, Langford HG, Oberman A, Jennings S, Hataway H, Stern J, Zimbaldi N. Trial of antihypertensive intervention and management: greater efficacy with weight reduction than with a sodium-potassium intervention. J Am Diet Assoc. 1993 Apr;93(4):408-15. doi: 10.1016/0002-8223(93)92286-7. PMID 8454808
- [Background] Davis BR, Oberman A, Blaufox MD, Wassertheil-Smoller S, Zimbaldi N, Kirchner K, Wylie-Rosett J, Langford HG. Lack of effectiveness of a low-sodium/high-potassium diet in reducing antihypertensive medication requirements in overweight persons with mild hypertension. TAIM Research Group. Trial of Antihypertensive Interventions and Management. Am J Hypertens. 1994 Oct;7(10 Pt 1):926-32. doi: 10.1093/ajh/7.10.926. PMID 7826557
- [Background] Wassertheil-Smoller S, Davis BR, Breuer B, Chang CJ, Oberman A, Blaufox MD. Differences in precision of dietary estimates among different population subgroups. Ann Epidemiol. 1993 Nov;3(6):619-28. doi: 10.1016/1047-2797(93)90085-i. PMID 7921310
- [Derived] Fretts AM, Follis JL, Nettleton JA, Lemaitre RN, Ngwa JS, Wojczynski MK, Kalafati IP, Varga TV, Frazier-Wood AC, Houston DK, Lahti J, Ericson U, van den Hooven EH, Mikkila V, Kiefte-de Jong JC, Mozaffarian D, Rice K, Renstrom F, North KE, McKeown NM, Feitosa MF, Kanoni S, Smith CE, Garcia ME, Tiainen AM, Sonestedt E, Manichaikul A, van Rooij FJ, Dimitriou M, Raitakari O, Pankow JS, Djousse L, Province MA, Hu FB, Lai CQ, Keller MF, Perala MM, Rotter JI, Hofman A, Graff M, Kahonen M, Mukamal K, Johansson I, Ordovas JM, Liu Y, Mannisto S, Uitterlinden AG, Deloukas P, Seppala I, Psaty BM, Cupples LA, Borecki IB, Franks PW, Arnett DK, Nalls MA, Eriksson JG, Orho-Melander M, Franco OH, Lehtimaki T, Dedoussis GV, Meigs JB, Siscovick DS. Consumption of meat is associated with higher fasting glucose and insulin concentrations regardless of glucose and insulin genetic risk scores: a meta-analysis of 50,345 Caucasians. Am J Clin Nutr. 2015 Nov;102(5):1266-78. doi: 10.3945/ajcn.114.101238. Epub 2015 Sep 9. PMID 26354543